CLINICAL TRIAL: NCT01332578
Title: A Comparison of Solid and Soluble Forms of Cold and Influenza Remedies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: C7591227
Record Dates: First submitted 2011-04-07; First posted 2011-04-11 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-04

CONDITIONS: Influenza; Common Cold
MeSH Terms: conditions — Influenza, Human; Common Cold | interventions — Acetaminophen; Phenylephrine; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Product (Experimental): Paracetamol, phenylephrine and ascorbic acid to be administered in 150 milliliters (mL) of hot water.
  Interventions: Drug: Paracetamol; Drug: Phenylephrine; Drug: Ascorbic Acid
- Paracetamol tablet (Active Comparator): Two paracetamol 500 mg tablets to be administered with 150 mL of hot water.
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Paracetamol — Present in both test and active comparator
Drug: Phenylephrine — Test product
  Arms: Test Product
Drug: Ascorbic Acid — Test product
  Arms: Test Product

SUMMARY:
The study is designed to investigate whether paracetamol from a hot remedy reaches the plasma faster than standard paracetamol tablets. The study will also assess the gastrointestinal transit of two oral cold and influenza ('flu') formulations using gamma scintigraphy. It is postulated that paracetamol in solution, such as from cold and 'flu' hot remedies, provides a greater early exposure compared to standard paracetamol tablets. In addition, the pharmacokinetic (PK) profile of paracetamol in the two formulations will be investigated.

ELIGIBILITY:
* Healthy male volunteers
* Body mass index between 18.0-29.9 kg/m^2

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- BIO-IMAGES Research Ltd., Glasgow, Scotland, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at one clinical study site in Glasgow.
Pre-assignment Details: Of 37 participants screened, 12 participants did not meet the study criteria. Remaining 25 participants were randomized into the study.
Groups:
- Hot Drink Remedy First, Then Standard Paracetamol Tablets: Participants received one sachet of hot drink remedy containing 1000 milligram (mg) paracetamol, 10 mg phenylephrine and 40 mg ascorbic acid in 150 milliliter (mL) of radio-labeled water (first intervention period). After a washout period of minimum two days, a single dose of two radio-labeled tablets of standard paracetamol (500 mg each) with 150 mL water were administered (second intervention period).
- Standard Paracetamol Tablets First, Then Hot Drink Remedy: Participants received a single dose of two radio-labeled tablets of standard paracetamol (500 mg each) with 150 mL of water (first intervention period). After a washout period of minimum two days, one sachet of hot drink remedy with 150 mL of radio-labeled water was administered (second intervention period).
Period: Period I
Arm/Group | Hot Drink Remedy First, Then Standard Paracetamol Tablets | Standard Paracetamol Tablets First, Then Hot Drink Remedy
Started | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | Hot Drink Remedy First, Then Standard Paracetamol Tablets | Standard Paracetamol Tablets First, Then Hot Drink Remedy
Started | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0
Period: Period II
Arm/Group | Hot Drink Remedy First, Then Standard Paracetamol Tablets | Standard Paracetamol Tablets First, Then Hot Drink Remedy
Started | 12 | 13
Completed | 12 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Randomized Participants: All randomized participants who received a study treatment during the cross over study.
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.5 (11.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Time to Reach Plasma Paracetamol Concentration of 0.25 μg/mL (Microgram Per Milliliter)
Description: Time to reach plasma paracetamol concentration of 0.25 μg/mL was determined using plasma concentration time profiles.
Time Frame: Blood samples taken within 15-30 minutes prior to dosing and at 3, 5, 7, 9, 11, 15, 20, 30, 45, 90, 120 and 180 minutes post-dose
Population: Modified Intent-To-Treat (MITT) population: all randomized participants with any post baseline pharmacokinetic measurement or scintigraphic measurement, and had evaluable data in at least one of the two study periods.
Measure: Median (Full Range); unit: minutes
Groups:
- Hot Drink Remedy: Participants received one sachet of hot drink remedy powder containing 1000 mg paracetamol, 10 mg phenylephrine and 40 mg ascorbic acid dissolved in 150 mL of radio-labeled water.
- Standard Paracetamol Tablets: Participants received a single dose of two radio-labeled tablets of standard paracetamol (500 mg each) with 150 mL of water.
Arm/Group | Hot Drink Remedy | Standard Paracetamol Tablets
Number analyzed (Participants) | 24 | 25
minutes | 4.59 [3.4 to 11.1] | 23.14 [6.0 to 46.6]
Statistical Analysis 1: Comparison: Hot Drink Remedy vs Standard Paracetamol Tablets; Null hypothesis was no difference between test hot drink and standard paracetamol tablets; Test type: Superiority or Other; p = 0.0004, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = -20.92, 95% CI 2-sided [-27.31 to -15.81] — Hodges-Lehmann estimate of median difference was determined

2. Secondary Outcome: Area Under the Concentration/Time Curve From 0 to 30 Minutes (Min) (AUC 0-30 Min)
Description: AUC (0-30 min) was determined from paracetamol plasma concentration time profiles using trapezoidal rule.
Time Frame: Blood samples taken within 15-30 min prior to dosing and at 3, 5, 7, 9, 11, 15, 20, 30, 45, 90, 120 and 180 minutes post-dose
Population: MITT population: all randomized participants with any post baseline pharmacokinetic measurement or scintigraphic measurement, and had evaluable data in at least one of the two study periods.
Measure: Mean (Standard Deviation); unit: nanograms (ng)*hours (h)/mL
Arm/Group | Hot Drink Remedy | Standard Paracetamol Tablets
Number analyzed (Participants) | 24 | 6
nanograms (ng)*hours (h)/mL | 1535.80 (873.300) | 387.28 (363.139)

3. Secondary Outcome: AUC (0-60 Min)
Description: AUC (0-60 min) was determined from paracetamol plasma concentration time profiles using trapezoidal method.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Hot Drink Remedy | Standard Paracetamol Tablets
Number analyzed (Participants) | 24 | 20
ng*h/mL | 5007.11 (1890.135) | 1874.22 (1555.539)

4. Secondary Outcome: Maximum Plasma Concentration (Cmax)
Description: Cmax was determined using plasma paracetamol concentration time profile.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Hot Drink Remedy | Standard Paracetamol Tablets
Number analyzed (Participants) | 24 | 25
ng/mL | 8309.58 (2109.196) | 9225.20 (1681.200)

5. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax)
Description: Time after administration when the maximum plasma concentration was reached.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Hot Drink Remedy | Standard Paracetamol Tablets
Number analyzed (Participants) | 24 | 25
hours | 1.50 [0.2 to 2.0] | 1.99 [0.7 to 3.0]

6. Secondary Outcome: Time to Onset of Gastric Emptying
Description: The individual anterior and posterior images were assessed using Gamma Scintigraphy images and WebLink Image Analysis program to determine the time to onset of gastric emptying of hot drink remedy and standard paracetamol tablets.
Time Frame: Baseline to 10 hours
Population: Period Level MITT population: all randomized participants with any post baseline pharmacokinetic measurement or scintigraphic measurement, and had evaluable data in one of the two study periods. Gastric emptying endpoints were only measured in the first period for each participant.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Hot Drink Remedy | Standard Paracetamol Tablets
Number analyzed (Participants) | 11 | 13
minutes | 7.86 (3.909) | 54.23 (3.596)

7. Secondary Outcome: Time to Completion of Gastric Emptying
Description: Time to completion of gastric emptying of hot drink remedy and standard paracetamol tablets was assessed using Gamma Scintigraphy images and WebLink image analysis program. Completion of gastric emptying was confirmed by two consecutive images with negligible gastric activity.
Time Frame: Baseline to 10 hours
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Hot Drink Remedy | Standard Paracetamol Tablets
Number analyzed (Participants) | 11 | 13
minutes | 202.59 (16.811) | 168.38 (15.463)

8. Secondary Outcome: Time to Onset and Completion of Disintegration of Reference Tablets
Description: Qualitative onset and completion of tablet disintegration was determined using Gamma scintigraphy images and WebLink image analysis program.
Time Frame: Baseline to 10 hours post dose
Population: Period Level MITT population: all randomized participants with any post baseline pharmacokinetic measurement or scintigraphic measurement, and had evaluable data in one of the two study periods. Tablet Disintegration endpoints were only measured in the first period for each participant.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Standard Paracetamol Tablets
Number analyzed (Participants) | 13
minutes
  Onset Time of Disintegration | 42.50 (18.028) [12.5 to 67.5]
  Completion Time of Disintegration | 62.88 (24.788) [22.5 to 112.5]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the start of the treatment, and until 5 days following administration of the last dose of investigational product.
Groups:
- Hot Drink Remedy: Participants then received one sachet of hot drink remedy powder containing 1000 mg paracetamol, 10 mg phenylephrine and 40 mg ascorbic acid, which was dissolved in 150 mL of radio-labeled water.
Arm/Group | Hot Drink Remedy | Standard Paracetamol Tablets
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 3/25 | 3/25
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hot Drink Remedy (N=25) | Standard Paracetamol Tablets (N=25)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Blood Bilirubin Increased (Investigations) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.